CLINICAL TRIAL: NCT07004712
Title: Efficacy and Biomarkers of the Second-line Treatment of Adebelizumab Combined With Irinotecan Liposome in Advanced Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Yang Wang, Associate Professor of Medicine, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCLC-001
Record Dates: First submitted 2025-05-13; First posted 2025-06-04 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; Adebelizumab combined with irinotecan liposome; second-line immnunotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): adebelizumab and irinotecan liposome
  Interventions: Drug: Adebelizumab combined with irinotecan liposome as second-line therapy

INTERVENTIONS:
Drug: Adebelizumab combined with irinotecan liposome as second-line therapy — Adebellizumab: intravenous drip, 1200mg, the infusion time is controlled between 30-60 minutes, and the infusion is completed within 2 hours at most. It is administered on the first day of each cycle and repeated once every 3 weeks.Irinotecan liposome: intravenous drip, 80mg/m2, infusion time of 30 minutes, the first dose of each cycle, repeated once every 3 weeks.After 4-6 cycles of adebelizumab combined with irinotecan liposome treatment, the subjects who did not develop the disease continued to use adebelizumab (1200mg, D1, Q3W) for maintenance treatment until the disease progressed, the toxicity was intolerable, the subjects voluntarily asked to withdraw and the researchers judged that the subjects needed to withdraw from the study.

SUMMARY:
This study is an open, single-arm, single-center phase II clinical study, which aims to evaluate the efficacy and safety of adebelizumab combined with irinotecan liposome in the second-line treatment of advanced small cell lung cancer, explore biomarkers to predict the efficacy, and further select the dominant population in immunotherapy.

In this study, 46 patients with extensive SCLC who had previously received immunotherapy combined with chemotherapy were enrolled. Subjects who met the enrollment conditions will be given adebelizumab combined with irinotecan liposome at the same time. After 4-6 cycles of treatment, if their condition has not progressed, they will be treated with adebelizumab until the disease progresses, toxicity can not be tolerated or other reasons specified in the scheme can be terminated. Subjects who finish the treatment will enter the follow-up period for safety follow-up and survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18-75 years old; 2. Small cell lung cancer diagnosed by histology; Compound small cell lung cancer is not allowed; 3. Progress in receiving first-line chemotherapy combined with immunotherapy (including PD-1 inhibitor and PD-L1 inhibitor); 4. According to RECIST 1.1 standard, there is at least one measurable objective lesion; 5.ECOG score 0-1; 6. The functions of important organs meet the following requirements:Bone marrow function: neutrophils ≥1.5×109/L, platelets ≥100×109/L, hemoglobin concentration ≥ 90g/L;Liver function: bilirubin ≤ 1.5× ULN; Aspartate aminotransferase and glutamate aminotransferase ≤2.5×ULN, and AST and ALT ≤ 5× ULN in case of liver metastasis; Total bilirubin ≤1.5 times the upper limit of normal value;Renal function: serum creatinine ≤1.5×ULN, or creatinine clearance rate (CCR) ≥ 60 ml/min; 7. Expected survival > 12 weeks;Patients have good compliance with the planned treatment, can understand the research process of this study and sign a written informed consent.

Exclusion Criteria:

1. Irinotecan liposome or Irinotecan has been used before; 2. Severe heart and lung diseases, new york Heart Association (NYHA) scores that patients with heart diseases above Grade II (including Grade II); 3. Patients with severe systemic infection or other serious diseases; 4. Patients who are known to be allergic or intolerant to chemotherapy drugs or their accessories; 5. Other malignant tumors have appeared in the past 5 years, except cured cervical carcinoma in situ and non-melanoma skin cancer; 6. Patients of childbearing age during pregnancy or lactation, and those who refused to take appropriate contraceptive measures during this experiment; 7. Have participated in clinical studies of other drugs within 21 days before the first dose of the study drug is given; 8. Combined with active autoimmune diseases and inflammatory diseases; 9. Grade 3-4 immune-related adverse reactions occurred during previous immunotherapy; 10. Symptomatic brain metastasis and meningeal metastasis; 11. Before the first administration, you are receiving long-term systemic corticosteroid therapy with prednisone > 10mg/d or equivalent anti-inflammatory active drugs or any form of immunosuppressive therapy. Subjects who need bronchodilators, inhaled or topical steroids or local steroid injections can be included in this study; 12. Patients with a large amount of serous cavity effusion, or serous cavity effusion with symptoms, or poor control of serous cavity effusion (poor control is defined as: puncture and drainage are needed twice or more in one month);The researcher judges the patients who are not suitable to participate in this study.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 0-12months
  It refers to the time from the date when the subjects enter the group to the time when the disease progresses or dies, whichever comes first.

SECONDARY OUTCOMES:
Percentage of Participants Who Had an Objective Response Rate(ORR) Based on Response Evaluation Criteria In Solid Tumors (RECIST) Criteria. | through study completion, an average of 1 year
  the proportion of subjects who achieve CR or PR as the best tumor remission during treatment.
Overall Survival (OS) | 0-5years
  The time from the date of admission to the death caused by any cause.
Safety: Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | through study completion, an average of 2 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Biomarker | "Baseline" and "after 2 cycles of treatment"
  ScRNA-seq was used to detect the puncture tissue samples before treatment, so as to analyze the influence of single cell level immune signal pathway and immune microenvironment on the efficacy of immunotherapy and explore biomarkers to predict the efficacy.
  At the same time, the peripheral blood samples were tested by metabonomics before treatment, after 2 cycles of evaluation and when the disease progressed, so as to explore metabolic markers that can predict and dynamically reflect the efficacy of immunotherapy through non-invasive liquid biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university cancer hospital, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: No